CLINICAL TRIAL: NCT03695536
Title: The Impact of Integration of Ultrasound on CPR Quality - A Video Review
Brief Title: The Impact of Integration of Ultrasound on CPR Quality - A Video Review Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807084RINB
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2018-09

CONDITIONS: Cardiopulmonary Resuscitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasound use during resuscitation: The group with ultrasound integrated into the resuscitation efforts.
  Interventions: Behavioral: ultrasound use during resuscitation
- no ultrasound use during resuscitation: The group without ultrasound integrated into the resuscitation efforts.

INTERVENTIONS:
Behavioral: ultrasound use during resuscitation — ultrasound use during resuscitation
  Groups: ultrasound use during resuscitation

SUMMARY:
High-quality cardiopulmonary resuscitation (CPR) is essential for return of spontaneous circulation (ROSC) in patients with cardiac arrest. However, some factors are known to be related with delays in chest compressions such as bed transfer, setting of CPR device, pulse and rhythm checks. This study aims to evaluate the potential impact of ultrasound on CPR quality by using retrospective video analysis.

All CPR scenarios in our department were recorded and masked for the purpose of video analysis. The investigators will record in-scene resuscitation manpower, the factors to interrupt chest compressions and whether introducing ultrasound into resuscitation process is related with delays in chest compressions. In addition, the investigators collect the patient's sex, age, initial rhythm and prognosis, including ROSC, survival to admission and survival to discharge.

ELIGIBILITY:
Inclusion Criteria:

adult patients (more than 20 years) non-traumatic cardiac arrest

Exclusion Criteria:

traumatic cardiac arrest age less than 20 years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (more than 20 years) with non-traumatic cardiac arrest at the emergency department of the National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Ultrasound use would not delay in chest compressions during resuscitation. | 60 minutes
  chest compression fraction (chest compression time/total resuscitation time) between two groups.

SECONDARY OUTCOMES:
Ultrasound use would not influence the rates of return of spontaneous circulation. | 60 mintues
  rates of return of spontaneous circulation.
Ultrasound use would not influence the rates of survival to admission. | 7 days.
  rates of survival to admision between two groups.
Ultrasound use would not influence the rates of survival to discharge. | 3 months.
  rates of survival to discharge between two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Department of Emergency Medicine, National Taiwan University Hospital, Taipei